CLINICAL TRIAL: NCT00960713
Title: The RITAI Cohort. An Observational Study on Serious Adverse Events Occuring After Rituximab Off-label Use for Auto-immune Disorders
Brief Title: The RITAI Cohort: An Observational Study on Rituximab Off-label Use for Auto-immune Disorders
Acronym: RITAI
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 0816002; AOL 2008
Record Dates: First submitted 2009-07-16; First posted 2009-08-18 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Pemphigus; Auto-immune Thrombocytopenic Purpura; Hemolytic Auto-immune Anaemia; Cold Agglutinin Disease; Cryoglobulinemia
Keywords: observational cohort; rituximab; off-label use; auto-immunity; cytopenia
MeSH Terms: conditions — Pemphigus; Anemia, Hemolytic, Autoimmune; Cryoglobulinemia; Cytopenia | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A biological collection will be constituted to allow pharmaco- immunological studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- The RITAI cohort: Every patient treated by rituximab off-label for auto-immune diseases in the public hospitals of the Midi-Pyrénées County (South of France) is eligible for the study, whatever the dose and planned infusions number. The enrolment is definitive when the first rituximab infusion begins. Follow-up visits are planned at months 1, 3, 6, 12 and 18 after the first infusion. At each visit, the investigators will record the adverse events that have occurred since the last visit. Serious or unexpected adverse events will be systematically monitored and declared to the Department of Pharmacology Pharmacovigilance unit and to Health Authorities (AFSSAPS). Imputability will be quoted according to the French method. A biological collection will be constituted to allow pharmaco-immunological studies.
  Interventions: Drug: Rituximab (MABTHERA® or RITUXAN®).

INTERVENTIONS:
Drug: Rituximab (MABTHERA® or RITUXAN®). — patients can be included in the study whatever the dosage used. Most patients will receive a classical 375 mg/m2 dose every week during four times (J0-J7-J14-J21).

SUMMARY:
The primary purpose of the study is to describe by a prospective observational study the serious adverse events occurring in patients treated off-label by rituximab for various auto-immune diseases.

DETAILED DESCRIPTION:
Every patient treated by rituximab off -label for auto-immune diseases in the public hospitals of the Midi-Pyrénées County (France) is eligible for the study, whatever the dose and the number of planned infusions. The enrollment is definitive at the time the first rituximab infusion begins. Follow-up visits are planned at months 1, 3, 6, 12 and 18 after the first infusion. At each visit, the investigators will record the adverse events that have occurred since the last visit. Serious or unexpected adverse events will be systematically monitored and declared to the Pharmacovigilance. Imputability will be quoted according to the French method. A biological collection will be constituted to allow pharmaco- immunological studies.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* rituximab is prescribed off-label for an auto-immune disorder
* rituximab prescription is validated by an institutional board
* Patients have given their informed consent to be included in the cohort

Exclusion Criteria:

* Follow-up for 6 months presumably doubtful
* Rituximab is prescribed for rheumatoïd arthritis
* Rituximab is prescribed for lymphoma
* Pregnant or breath feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient treated by rituximab off -label for auto-immune diseases in the public hospitals of the Midi-Pyrénées County (in the South of France) is eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of a serious adverse events | Day 14, Week 6, Month 6, Month 12 and Month 18

SECONDARY OUTCOMES:
Type, severity and frequency of all other adverse events occurring in the year following rituximab | Day 14, Week 6, Month 6, Month 12 and Month 18
Factors that may influence the occurrence of infectious adverse events | Day 14, Week 6, Month 6, Month 12 and Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Sailler, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de médecine interne, hôpital Purpan, place du Dr Baylac, Toulouse, France